CLINICAL TRIAL: NCT04914247
Title: Individual Patient Expanded Access IND for Selexipag (Uptravi) in Participants With Non-healing Wound, Buerger's Disease
Status: Available | Type: Expanded Access
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108669; 67896049PAH4002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Non-healing Wound; Thromboangiitis Obliterans
MeSH Terms: conditions — Thromboangiitis Obliterans | interventions — selexipag

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Selexipag

SUMMARY:
The purpose of this expanded access program (EAP) is to provide Selexipag (Uptravi) for the treatment of participant with non-healing wound, buerger's disease.

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion